CLINICAL TRIAL: NCT00111306
Title: A Phase III, Randomized, Double-Blind. Placebo-Controlled, Multi-Center Study of Systemic Lupus Erythematosus With Acute Severe SLE Flares Excluding Renal or Neurological Systems
Brief Title: Study of Epratuzumab in Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL0003 (IMMU-103-03); EudraCT #: 2005-000705-59
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Antibody; B-cell immunotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

INTERVENTIONS:
Drug: epratuzumab

SUMMARY:
The purpose of the study is to evaluate the safety & efficacy of Epratuzumab with standard treatments for patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Has SLE by ACR revised criteria (meets <4 criteria);
* Has SLE with at least one elevated lupus antibody;
* Has new onset of severe lupus disease flare in at least one body or organ system, excluding renal or neurologic

Exclusion Criteria:

* Active severe CNS or Renal disease defined by BILAG as Level A
* Allergy to murine or human antibodies
* Antiphospholid antibodies AND a history of thrombocytopenic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510
Dates: Start 2005-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Patient response variable (complete response, partial response, non-response) evaluated at 24 weeks.

SECONDARY OUTCOMES:
Proportion of patients with complete response or partial response;
Individual BILAG assessments;
Physician and patient assessment scores;
Time-to treatment failure;
Successful steroid reduction by weeks 20 and 24;
Maintenance of steroid reduction at 24 and 48 weeks;
Monitor the plasma concentration and immunogenicity profile of epratuzumab in patients with Lupus;
Assess epratuzumab on Health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Barry, Study Director — UCB Pharma
Locations (18):
- United States (13):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Upland, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Baltimore, Maryland
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Charleston, South Carolina
- Brussels, Belgium
- Debrecen, Hungary
- Amsterdam, Netherlands
- Santander, Spain
- Birmingham, United Kingdom

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069